CLINICAL TRIAL: NCT00004026
Title: A Phase II Study of CT-2584 Mesylate in Patients With Hormone Refractory Prostate Cancer
Brief Title: CT-2584 in Treating Patients With Metastatic Prostate Cancer That Has Not Responded to Previous Therapy
Status: Terminated | Phase: Phase 2 | Type: Interventional
Sponsor: CTI BioPharma (Industry)
Allocation: Randomized | Purpose: Treatment
Other Study IDs: CTI-1038; CDR0000067257 (Registry Identifier: PDQ (Physician Data Query)); CPMC-IRB-8781
Record Dates: First submitted 1999-11-01; First posted 2004-08-27 (Estimated); Last update posted 2020-10-19 (Actual); Status verified 2020-10

CONDITIONS: Prostate Cancer
Keywords: adenocarcinoma of the prostate; stage IV prostate cancer; recurrent prostate cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — CT 2584; Drug Therapy

INTERVENTIONS:
Drug: CT-2584
Drug: chemotherapy

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. CT-2584 may stop the growth of prostate cancer by stopping blood flow to the tumor.

PURPOSE: Randomized phase II trial to study the effectiveness of CT-2584 in treating patients who have metastatic prostate cancer that has not responded to previous therapy.

DETAILED DESCRIPTION:
OBJECTIVES: I. Compare the efficacy, safety, and pharmacokinetics of 2 different treatment schedules of CT-2584 in patients with hormone refractory, metastatic adenocarcinoma of the prostate.

OUTLINE: This is a randomized, multicenter study. Patients are randomized to 1 of 2 treatment arms: Arm I: Patients receive CT-2584 IV over 6 hours daily for 3 days every 3 weeks. Arm II: Patients receive CT-2584 IV over 6 hours once every 7 days for 3 weeks. Courses repeat every 3 weeks in the absence of disease progression or unacceptable toxicity.

PROJECTED ACCRUAL: Approximately 80 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Histologically proven metastatic adenocarcinoma of the prostate Refractory to hormonal therapy Failed at least 1 nonhormonal therapy (prior radiotherapy allowed, but does not constitute nonhormonal therapy) No CNS metastases

PATIENT CHARACTERISTICS: Age: 18 and over Performance status: 60-100% Life expectancy: Not specified Hematopoietic: No known or suspected red blood cell disorder (e.g., hereditary spherocytosis, paroxysmal nocturnal hematuria, sickle cell trait, autoimmune hemolytic disorder) Hepatic: Bilirubin no greater than 1.5 mg/dL No severe liver dysfunction, particularly, no impaired hepatic synthetic functions as evidenced by prolonged prothrombin time or otherwise unexplained serum albumin less than 3 g/dL Renal: Creatinine no greater than 1.5 mg/dL Cardiovascular: No evidence of congestive heart failure No clinically significant cardiac arrhythmia No prior or concurrent symptoms of acute coronary artery disease No significant cardiac valve disease (e.g., aortic stenosis, valve prosthesis) Pulmonary: No prior asthma during adulthood that required therapy Other: No prior seizures or drug related anaphylactic reactions No history of microangiopathy (e.g., cavenous hemangioma, prior thrombotic thrombocytopenic purpura)

PRIOR CONCURRENT THERAPY: Biologic therapy: At least 4 weeks since prior systemic biologic therapy for prostate cancer and recovered Chemotherapy: At least 4 weeks since prior chemotherapy (12 weeks for strontium-89 and 6 weeks for bicalutamide) and recovered Endocrine therapy: See Disease Characteristics Radiotherapy: See Disease Characteristics No concurrent radiotherapy Surgery: At least 3 weeks since prior major thoracic or abdominal surgery Other: At least 4 weeks since other prior investigational drugs (except bisphosphonates) and recovered

Ages: 18 Years to 120 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 1998-12 (Actual); Primary Completion 2005-01 (Actual); Study Completion 2005-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Carolyn Paradise, MD, Study Chair — CTI BioPharma
Locations (7):
- United States (7):
  - Jonsson Comprehensive Cancer Center, UCLA, Los Angeles, California
  - UCSF Cancer Center and Cancer Research Institute, San Francisco, California
  - Stanley Scott Cancer Center, New Orleans, Louisiana
  - Johns Hopkins Oncology Center, Baltimore, Maryland
  - Herbert Irving Comprehensive Cancer Center, New York, New York
  - Our Lady of Mercy Medical Center, The Bronx, New York
  - University of Washington Medical Center, Seattle, Washington